CLINICAL TRIAL: NCT06582940
Title: Elimination of PTV Margins Based on MRI-guided Adaptive Stereotactic Radiotherapy for Non-small Cell Lung Cancer With Brain Metastasis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Liu, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GASTO-10115
Record Dates: First submitted 2024-08-28; First posted 2024-09-03 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: MRI-guided Adaptive Radiotherapy; Non-small Cell Lung Cancer; Brain Metastasis
Keywords: MRI-guided radiotherapy; lung cancer; brain metastasis
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms; Lung Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The study group (Experimental): Patients in the study group will receive MRI-guided adaptive stereotactic radiotherapy (without PTV expansion margin). The total dose will be 30Gy/5 fractions, administered once daily. The MRI-linac is used for the delivery of radiotherapy.
  Interventions: Radiation: MRI-guided adaptive SRT
- The control group (Active Comparator): Patients in the study group will receive conventional standard stereotactic radiotherapy (with PTV expansion margin). The total dose will be 30Gy/5 fractions, administered once daily. The conventional linac is used for the delivery of radiotherapy.
  Interventions: Radiation: Conventional SRT

INTERVENTIONS:
Radiation: MRI-guided adaptive SRT — MRI-guided online adaptive SRT (without PTV expansion margin). The total dose will be 30Gy/5 fractions, administered once daily. MRI will be acquired.
  Arms: The study group
Radiation: Conventional SRT — Conventional SRT (with PTV expansion margin). The total dose will be 30Gy/5 fractions, administered once daily. CBCT will be acquired.
  Arms: The control group

SUMMARY:
This study aims to explore the safety and efficacy of eliminating the planning target volume (PTV) margins based on MRI-guided adaptive stereotactic radiotherapy for non-small cell lung cancer (NSCLC) patients with brain metastasis.

DETAILED DESCRIPTION:
This study aims to explore the safety and efficacy of eliminating the planning target volume (PTV) margins based on MRI-guided adaptive stereotactic radiotherapy for NSCLC patients with brain metastasis. In this study, patients will be randomly assigned in a 1:1 ratio to the study group or the control group. Patients in the study group will receive MRI-guided adaptive stereotactic radiotherapy (SRT) (without PTV expansion margin), while patients in the control group will receive CT-guided conventional standard SRT (with PTV expansion margin). After the completion of treatment, patients will be followed up regularly to assess safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years
* Histologically or cytologically confirmed non-small cell lung cancer
* 1-10 metastases on contrast-enhanced MRI
* Radiotherapy for extracranial lesions is permitted
* Tyrosine kinase inhibitors (TKI) are permitted in patients with progression of
* intracranial metastases during previous TKI therapy
* Patients have measurable or evaluable lesions based on the Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Normal function of organs and bone marrow within 14 days: Total bilirubin 1.5 times or less the upper limits of normal (ULN); AST and ALT 1.5 times or less the ULN; absolute neutrophil count≥ 500 cells/mm3; creatinine clearance rate(CCR) ≥45 mL/min; Platelet count≥50,000 cells/mm3; international normalized ratio(INR) ≤1.5#Prothrombin Time (PT)≤ 1.5 × ULN
* Informed-consent

Exclusion Criteria:

* Small cell carcinoma of lung
* Intracranial metastases needed surgical decompression
* Patients with contraindications for MRI
* Previous radiotherapy or excision for intracranial metastases
* Hypertensive crisis, hypertensive encephalopathy, symptomatic heart failure (New York class II or above), active cerebrovascular disease or cardiovascular disease occurred within 6 months
* Uncontrolled hypertension (systolic > 150mmHg and/or diastolic > 100mmHg)
* Major surgery within 28 days or minor surgery or needle biopsy within 48 hours
* Urine protein 3-4+, or 24h urine protein quantitative >1g
* Severe uncontrolled disease
* Uncontrollable seizure or psychotic patients without self-control ability
* Women in pregnancy, lactation period
* Other not suitable conditions determined by the investigators

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Radiation-related brain necrosis incidence rate | 1 year
  "Radiation-related brain necrosis" refers to brain tissue damage that occurs as a result of radiation therapy. It can be detected by brain MRI imaging.

SECONDARY OUTCOMES:
intracranial progression-free survival rate | 1 year
  The percentage of patients who, after one year of treatment, have not experienced any progression of their intracranial disease.
Objective response rate | 1-year
  To evaluate the effectiveness of a treatment for brain tumors based on RECIST 1.1 criteria.
Overall survival | 1 year
  The percentage of patients who are alive after one year of treatment.
Radiation-related Neurotoxicity | 1 year
  "Neurotoxicity" refers to the harmful effects that certain substances or conditions can have on the nervous system, which was examined based on RECIST 1.1 criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shaw MG, Ball DL. Treatment of brain metastases in lung cancer: strategies to avoid/reduce late complications of whole brain radiation therapy. Curr Treat Options Oncol. 2013 Dec;14(4):553-67. doi: 10.1007/s11864-013-0258-0. PMID 24048959
- [Background] Baliga S, Garg MK, Fox J, Kalnicki S, Lasala PA, Welch MR, Tome WA, Ohri N. Fractionated stereotactic radiation therapy for brain metastases: a systematic review with tumour control probability modelling. Br J Radiol. 2017 Feb;90(1070):20160666. doi: 10.1259/bjr.20160666. Epub 2016 Dec 12. PMID 27936894
- [Background] Lagendijk JJ, Raaymakers BW, Van den Berg CA, Moerland MA, Philippens ME, van Vulpen M. MR guidance in radiotherapy. Phys Med Biol. 2014 Nov 7;59(21):R349-69. doi: 10.1088/0031-9155/59/21/R349. Epub 2014 Oct 16. No abstract available. PMID 25322150
- [Background] Khoo VS, Joon DL. New developments in MRI for target volume delineation in radiotherapy. Br J Radiol. 2006 Sep;79 Spec No 1:S2-15. doi: 10.1259/bjr/41321492. PMID 16980682
- [Background] Stemkens B, Tijssen RH, de Senneville BD, Lagendijk JJ, van den Berg CA. Image-driven, model-based 3D abdominal motion estimation for MR-guided radiotherapy. Phys Med Biol. 2016 Jul 21;61(14):5335-55. doi: 10.1088/0031-9155/61/14/5335. Epub 2016 Jun 30. PMID 27362636
- [Background] Glitzner M, Crijns SP, de Senneville BD, Kontaxis C, Prins FM, Lagendijk JJ, Raaymakers BW. On-line MR imaging for dose validation of abdominal radiotherapy. Phys Med Biol. 2015 Nov 21;60(22):8869-83. doi: 10.1088/0031-9155/60/22/8869. Epub 2015 Nov 4. PMID 26531846
- [Background] Ma LH, Li G, Zhang HW, Wang ZY, Dang J, Zhang S, Yao L, Zhang XM. Hypofractionated stereotactic radiotherapy with or without whole-brain radiotherapy for patients with newly diagnosed brain metastases from non-small cell lung cancer. J Neurosurg. 2012 Dec;117 Suppl:49-56. doi: 10.3171/2012.7.GKS121071. PMID 23205789
- [Background] Raaymakers BW, Jurgenliemk-Schulz IM, Bol GH, Glitzner M, Kotte ANTJ, van Asselen B, de Boer JCJ, Bluemink JJ, Hackett SL, Moerland MA, Woodings SJ, Wolthaus JWH, van Zijp HM, Philippens MEP, Tijssen R, Kok JGM, de Groot-van Breugel EN, Kiekebosch I, Meijers LTC, Nomden CN, Sikkes GG, Doornaert PAH, Eppinga WSC, Kasperts N, Kerkmeijer LGW, Tersteeg JHA, Brown KJ, Pais B, Woodhead P, Lagendijk JJW. First patients treated with a 1.5 T MRI-Linac: clinical proof of concept of a high-precision, high-field MRI guided radiotherapy treatment. Phys Med Biol. 2017 Nov 14;62(23):L41-L50. doi: 10.1088/1361-6560/aa9517. PMID 29135471